CLINICAL TRIAL: NCT04579367
Title: Non-interventional Study on the Treatment With Bempedoic Acid and/or Its Fixed-dose Combination With Ezetimibe in Routine Clinical Practice in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia (MILOS)
Brief Title: Treatment With Bempedoic Acid and/or Its Fixed-dose Combination With Ezetimibe in Primary Hypercholesterolemia or Mixed Dyslipidemia
Acronym: MILOS
Status: Active, not recruiting | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DSE-BMP-01-20-EU
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Hypercholesterolemia; Mixed dyslipidemia; Bempedoic acid and/or its fixed-dose combination with ezetimibe
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bempedoic acid and/or fixed-dose combination with ezetimibe: Participants with primary hypercholesterolemia or mixed dyslipidemia who received bempedoic acid and/or its fixed-dose combination with ezetimibe.
  Interventions: Drug: Bempedoic acid and/or its fixed-dose combination with ezetimibe

INTERVENTIONS:
Drug: Bempedoic acid and/or its fixed-dose combination with ezetimibe — This is a non-interventional study. No study medication will be provided to the patients. Medication will be prescribed by the treating physician in line with the clinical practice.

SUMMARY:
The primary objective is to describe in the real-world setting patient characteristics and outcomes of patients with primary hypercholesterolaemia (heterozygous familial and non-familial) or mixed dyslipidaemia using bempedoic acid and/or its fixed-dose combination with ezetimibe in managing plasma levels of low-density lipoprotein cholesterol (LDL-C).

Secondary objectives are to document and evaluate as applicable:

* Assessment of the cardiovascular risk of patients treated with bempedoic acid and/or its fixed-dose combination with ezetimibe using different risk scores (e.g. Systematic Coronary Risk Estimation (SCORE) system, SMART score for Very High Risk patients and Framingham risk score for High Risk patients. The scores will be re-calculated during the analysis and used as an analytical tool only).
* Changes in low-density lipoprotein cholesterol (LDL-C) levels prior to treatment with bempedoic acid and/or its fixed-dose combination with ezetimibe compared to 1 year follow-up and subsequent data collection points, if applicable.
* Characterize plasma levels of other potentially ASCVD-modifying cholesterol fragments, namely, LDL-C, total cholesterol (TC), apolipoprotein B (apoB), high-density lipoprotein cholesterol (HDL-C), non-HDL-C, triglycerides (TGs) and lipoprotein A (Lp[a]) compared to 1 year follow-up and subsequent data collection points, if applicable.
* Changes in the levels of inflammatory marker hsCRP compared to 1 year follow-up and subsequent data collection points, if applicable.
* Adverse Drug Reactions associated to bempedoic acid and/or its fixed-dose combination with ezetimibe.
* Changes in uric acid levels compared to 1 year follow-up and subsequent data collection points, if applicable.
* Relevant CV events:

  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery (CABG)
  * Percutaneous transluminal coronary angioplasty (PTCA)
  * Stroke
  * Transient ischemic attack (TIA)
  * Acute peripheral arterial occlusion
  * All-cause death
  * Cardiovascular (CV)-death
* Adverse effects associated with lipid-modifying treatment (LMT)

  * Laboratory abnormalities
  * Muscle-associated symptoms
  * New onset and/or worsening diabetes
  * Changes in the patients´ glycemic status over time
* Site characteristics (sites and practitioners) caring for patients treated with bempedoic acid and/or its fixed-dose combination with ezetimibe.
* Use of LMTs prior or concomitantly to receiving bempedoic acid and/or its fixed-dose combination with ezetimibe (therapies including combination treatments).
* Bempedoic acid and/or its fixed-dose combination with ezetimibe treatment parameters such as treatment duration by therapy, dosage, prescription intervals, permanent discontinuations, switches and reasons for these, (concomitant medication, additional therapy/interventions).
* Healthcare resource use especially consultation visits with specialist, nurse time and hospitalizations as well as patient-reported outcome using EQ-5D-5L and PAM-13.

DETAILED DESCRIPTION:
This non-interventional study will be conducted to characterize the risks and benefits of bempedoic acid and/or its fixed-dose combination with ezetimibe in a real-world clinical setting in adult patients with primary hypercholesterolaemia or mixed dyslipidaemia and to gain insight into the effectiveness (managing plasma levels of low-density lipoprotein cholesterol) as well as safety (clinical events associated with the treatment modalities). Real world evidence will be collected in 5000 participants, treated by specialized as well as non-specialized physicians in hospitals and office based centers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate
* At least 18 years of age
* Participants suffering from documented primary hypercholesterolemia or mixed dyslipidemia treated or intended to be treated with bempedoic acid and/or its fixed dose combination with ezetimibe at the discretion of the physician are appropriate for participation in the observation.
* No contraindications exist according to the SmPC of bempedoic acid and/or its fixed-dose combination with ezetimibe
* No concurrent participation in an interventional study (simultaneous participation in other non-interventional study is possible)
* Life expectancy > 1 year

Exclusion Criteria:

* As this is a non-interventional study, no explicit exclusion criteria are defined. The prescribing behavior will not be influenced. Only patients will be included where the decision has been made by the treating physician to treat the patients either with bempedoic acid and/or its fixed-dose combination with ezetimibe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with primary hypercholesterolemia or mixed dyslipidemia who are being treated with bempedoic acid and/or its fixed dose combination with ezetimibe.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Summary of patient characteristics in patients with primary hypercholesterolemia or mixed dyslipidemia following treatment with bempedoic acid and/or its fixed-dose combination with ezetimibe | Baseline (date of signed informed consent) up to 1 year minimum or 2 year maximum follow up (depending on the availability of bempedoic acid in countries)

SECONDARY OUTCOMES:
Overview of the cardiovascular risk of patients with primary hypercholesterolemia or mixed dyslipidemia following treatment with bempedoic acid/ and/or its fixed-dose combination with ezetimibe | Baseline (date of signed informed consent) up to 1 year minimum or 2 year maximum follow up (depending on the availability of bempedoic acid in countries)
  Cardiovascular risk scores will be assessed using the Systematic Coronary Risk Estimation (SCORE) system, Second manifestations of arterial disease (SMART) and Framingham risk scores. The SMART risk score will estimate 10-year risk for very high-risk participants based on clinical patient characteristics. The gender-specific Framingham risk score will be used to estimate 10-year cardiovascular risk for high-risk participants.
Summary of changes in plasma low-density lipoprotein cholesterol levels following treatment with bempedoic acid and/or its fixed-dose combination with ezetimibe in patients with primary hypercholesterolemia or mixed dyslipidemia | Baseline (date of signed informed consent) up to 1 year minimum or 2 year maximum follow up (depending on the availability of bempedoic acid in countries)
Summary in changes in plasma levels of atherosclerotic cardiovascular disease-modifying cholesterol fragments following treatment with bempedoic acid and/or its fixed-dose combination with ezetimibe | Baseline (date of signed informed consent) up to 1 year minimum or 2 year maximum follow up (depending on the availability of bempedoic acid in countries)
  Plasma levels of total cholesterol (TC), apolipoprotein B (apoB), high-density lipoprotein cholesterol (HDL-C), triglycerides (TGs) and lipoprotein a (Lp[a]) will be assessed.
Summary of changes in plasma inflammatory marker hsCRP levels following treatment with bempedoic acid and/or its fixed-dose combination with ezetimibe in patients with primary hypercholesterolemia or mixed dyslipidemia | Baseline (date of signed informed consent) up to 1 year minimum or 2 year maximum follow up (depending on the availability of bempedoic acid in countries)
  Inflammatory status was assessed using high-sensitive C-reactive protein.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company
Locations (444):
- Austria (20):
  - Dr. Armin Öhlinger Kardiologe & innere Medizin, Dornbirn
  - Landeskrankenhaus Feldkirch, Feldkirch
  - LKH-Univ. Klinikum Graz, Graz
  - Medizinische Universität Graz, Graz
  - Internist Dr. med. univ. Stefan Moser, Hörsching
  - Medizinische Universität Innsbruck, Innsbruck
  - KABEG Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Ordination Dr. Johannes Föchterle, Linz
  - Ordination Frau Prof. Dr. Yvonne Winhofer-Stöckl, Mattersburg
  - Kompetenz-Zentrum Diabetes, Salzburg
  - Ordination Universitätsdozent Dr. Alexander Kober, Sankt Aegyd am Neuwalde
  - Ordination Dr. med. univ. Evelyn Fließer-Görzer, Sankt Stefan ob Stainz
  - Ordination Dr. Thomas Maca, Vienna
  - Klinik Hietzing, Wiener Gesundheitsverbund, Vienna
  - Zentrum für Klinische Studien Dr. Hanusch GmbH, Vienna
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Univ.-Prof. Dr. Thomas Stulnig, Vienna
  - Herz Zentrum Währing, Vienna
  - Karl Landsteiner Institut für kardiovaskuläre und intensivmedizinische Forschung, Vienna
- Belgium (36):
  - ASZ, Aalst
  - Clinique Saint-Luc Bouge Namur, Bouge
  - Epicura Hornu, Boussu
  - A.Z. KLINA Brasschaat, Brasschaat
  - Clinique Saint-Jean Bruxelles, Brussels
  - CHU Brugman, Brussels
  - CUB-Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Clinique de l'Europe Saint Elisabeth, Brussels
  - UCL Saint-Luc Woluwé Bruxelles, Brussels
  - Private Practice, Ciney
  - Az Sint Blazius, Dendermonde
  - UZ Antwerpen, Edegem
  - Z.O.L - Campus St. Jan, Genk
  - AZ St-Lucas & Volkskliniek, Ghent
  - UZ Gent, Ghent
  - GHDC Charleroi - Site Hôpital Saint-Joseph, Gilly
  - Private Practice, Gribomont
  - Pôle hospitalier Jolimont, Haine-Saint-Paul
  - BVBA Med Kab, Halen
  - Jessa Ziekenhuis, Hasselt
  - CHR Huy, Huy
  - JAN YPERMAN Ziekenhuis, Ieper
  - AZ Groeninge Kortrijk, Kortrijk
  - CHU Tivoli, La Louvière
  - UZ Leuven, Leuven
  - CHR Citadelle de Liège, Liège
  - CHU Liège, Liège
  - CHU Charleroi Hopital civil Marie-Curie, Lodelinsart
  - CHU Mons Ambroise Paré, Mons
  - AZ Sint Jan, Ostend
  - AZ Delta, Roeselare
  - AZ Glorieux, Ronse
  - Sint Trudo, Sint-Truiden
  - Sint-Andriesziekenhuis Tielt, Tielt
  - CHU UCL Mont-Godinne, Yvoir
- Germany (147):
  - Downtown Clinic Aachen, Aachen
  - Praxis Delonge, Aachen
  - Praxis Osterziel, Amberg
  - MVZ Helios Aue, Aue
  - Kardiologische Praxis Enders, Bad Elster
  - SLK-Klinikum am Plattenwald, Bad Friedrichshall
  - Herzcarre Praxis, Bad Homburg
  - Kardiologische Praxis, Bad Homburg
  - Zentrum für klinische Forschung, Bad Homburg
  - Universitätsklinikum Freiburg - Universitäts-Herzzentrum, Bad Krozingen
  - Praxis am Landratspark, Bad Segeberg
  - Hausärzte am Spritzenhaus, Baiersbronn
  - CIMS Studienzentrum Bamberg GmbH Drs. Kirschner/Haas/Ritzel, Bamberg
  - Kardiologische Praxis, Bechhofen
  - Praxis Rankestraße, Berlin
  - SKP Studienzentrum der kardiologischen Praxisgemeinschaft Rankestrasse GmbH, Berlin
  - Herzpraxis Berlin MVZ, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Dres. Seeger & Partner, Berlin
  - Diabetespraxis Dr. Braun, Berlin
  - Lipidambulanz Charite, Berlin
  - Praxiszentrum Biedenkopf, Biedenkopf
  - Praxis Dr. A. Biedermann, Blankenhain
  - Kardiologische Gemeinschaftspraxis Bremerhaven, Bremerhaven
  - Kardiologie im Friedrichspalast Bruchsal, Bruchsal
  - MediClin Reha-Zentrum Spreewald, Burg
  - Studiengesellschaft Könemann und Steinmann GbR, Bünde
  - MVZ am Küchwald, Chemnitz
  - Kardiologische Praxis Stellmach, Chemnitz
  - MVZ Polymed, Chemnitz
  - Uniklinik Köln, Cologne
  - Zentrum für klinische Forschung, Cologne
  - IKAPP, Cologne
  - Praxis Dr. Menzel, Dessau
  - Klinikum Lippe GmbH, Detmold
  - Kardiologische Gemeinschaftspraxis, Dortmund
  - Cardiologicum Dresden/Pirna, Dresden
  - Hausärztliche Gemeinschaftspraxis mit diabetologischem Schwerpunkt, Dresden
  - Dres. Günther/Kolschmann, Dresden
  - Herzzentrum Dresden, Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - DZDM Diabeteszentrum Duisburg Mitte, Duisburg
  - Nierenzentrum Düren, Düren
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Praxis Dilltal, Ehringshausen
  - Praxis Dipl. -Med. Petra Herrmann, Eisenach
  - Kardiologische Praxis, Elsterwerda
  - Gemeinschaftspraxis ISP Erlangen, Erlangen
  - Hausarztzentrum am Germaniaplatz, Essen
  - DIAKO Flensburg, Flensburg
  - Praxis für Nieren und Hochdruck-Krankheiten, Flensburg
  - MVZ Altstadt-Carree Fulda, Fulda
  - Klinikum Fulda, Fulda
  - Praxis Dr. Langel, Gera
  - Cardiocampus Gemeinschaftspraxis für Herz- und Kreislauferkrankungen, Gifhorn
  - Praxis für Gefäßmedizin, Görlitz
  - Universitätsmedizin Göttingen, Göttingen
  - Praxis Dr. Müller, Gräfenhainichen
  - Universitätsmedizin Greifswald, Greifswald
  - Evangelisches Krankenhaus Hagen-Haspe, Hagen
  - Praxis, Hainburg
  - Cardiologicum Hamburg - Praxis Wandsbek, Hamburg
  - Diabetes Zentrum Wandsbeck, Hamburg
  - MVZ Prof. Mathey, Prof. Schofer, Hamburg
  - Kardiologie am Tibarg, Hamburg
  - Kardiologie List, Hanover
  - Kardiologische Praxis, Hanover
  - Kardiologische Praxis, Haßloch
  - Kardiologische Schwerpunktpraxis, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Praxis Heik/Wedig, Heiligenstadt
  - KARDIO-IN Kardiologische Gemeinschaftspraxis, Ingolstadt
  - Kardiologische Praxis, Kaiserslautern
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad
  - B. Braun Ambulantes Herzzentrum Kassel, Kassel
  - Praxis Dr. Heiner Müller, Katzhütte
  - Nephrologie Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein, Koblenz
  - Studienzentrum der Inneren Medizin I & II am Klinikum Konstanz, Konstanz
  - Kardiologie Dr. med. E. Persicke / Dr. med. O. Scheuermann, Kornwestheim
  - Kardiologische Praxis Kyritz, Kyritz
  - Universitätsklinikum Leipzig, Leipzig
  - Kardiologische Praxis Boudriot, Leipzig
  - MVZ Stoffwechselmedizin Leipzig, Leipzig
  - Praxis Dr. I.Simon-Wagner, Lichtenfels
  - St. Vincenz Krankenhaus, Limburg
  - Gemeinschaftspraxis Dr. Jens Biesenbaum und Dr. Uwe Gerbaulet, Löhne
  - Cardio Centrum Ludwigsburg-Bietigheim, Ludwigsburg
  - Kardiologische Praxisklinik Ludwigshafen, Ludwigshafen
  - Universität zu Lübeck, Lübeck
  - Institut für Präventive Medizin & Klinische Forschung GbR, Magdeburg
  - Cardiopraxis Mainz, Mainz
  - Katholisches Klinikum Mainz, Mainz
  - Universitätsklinikum Mainz, Mainz
  - ZE:RO Praxen, Mannheim
  - UMM Mannheim, Mannheim
  - Kardiologische Praxis, Markkleeberg
  - Praxis Ben-Chur, Meiningen
  - Praxis Haj-Yehia, Moers
  - Gemeinschaftspraxis Dr. Prohaska/Dr. Schulte, Mühldorf
  - Kardiologie Mühldorf am Inn, Mühldorf
  - Herzquartier Mülheim, Mülheim
  - Kardiologie Neuhausen-Nymphenburg, München
  - Dres. Wauer/Windstetter, München
  - Praxis Kiepenkerl, Münster
  - Zentrum für Kardiologie an der Raphaelsklinik Münster, Münster
  - Praxis für Innere Medizin Münster, Münster
  - Universitätsklinikum Münster, Münster
  - Internistische Praxisgemeinschaft, Neu-Isenburg
  - Kardiologische Praxis Northeim, Northeim
  - Hausarztpraxis, Oer-Erkenschwick
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Kardiologische Praxis Papenburg - Site 6071, Papenburg
  - Kardiologische Praxis Papenburg - Site 6072, Papenburg
  - Gemeinschaftspraxis Dres. med. Karl-Heinz Göttl - Omar Adjan, Passau
  - Hausärztlich-Kardiologisches MVZ "Am Felsenkeller" GmbH, Pirna
  - Kinikum Ernst von Bergmann, Potsdam
  - VieSante Herzmedizin Potsdam, Potsdam
  - Kardiologische Gemeinschaftspraxis, Potsdam
  - Allgemeinmedizinisch Internistische Praxis Dr. H. Borgmann, Radebeul
  - Internistisch hausärtzliche Gemeinschaftspraxis Dr. Hildebrandt & Dr. Mutscher, Radebeul
  - Gemeinschaftspraxis Herz Riesa, Riesa
  - Universitätsmedizin Rostock, Rostock
  - Facharztpraxis für Kardiologie und Innere Medizin, Schwäbisch Hall
  - MVZ Schwerin West GmbH, Schwerin
  - Nierenzentrum Altmark, Seehausen
  - Zentrum für Prävention und Rehabilitation, Siegen
  - Klinik Singen, Singen
  - MEDINOS Klinik Sonneberg, Sonneberg
  - Kardiologische Praxis im Steiner Thor, Straubing
  - Praxis Dr Knöbel u. Partner, Straubing
  - Praxis Dr. Michael Rother, Strausberg
  - Diabetologische Schwerpunktpraxis, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Studienzentrum der Herzklinik Ulm GbR, Ulm
  - Praxis Dr. Hansen, Unterwellenborn
  - Praxis Dr. Dengler/Hohenstatt, Ursensollen
  - Herzzentrum Saar, Völklingen
  - GRN Weinheim, Weinheim
  - Kardiologische Praxis Al-Zoebi, Wermsdorf
  - Internistische Gemeinschaftspraxis Dr. med. Schreckenberg, Dr. med. Vorderstraße, Weyhe
  - Forschungszentrum-Ruhr / KliFoCenter GmbH, Witten
  - Kardiologische Praxis Tamm/Hoh, Wittenberg
  - Kardiologische Fachpraxis, Wolmirstedt
  - Zentrum für Nieren- und Hochdrucklerkrankungen Hofaue, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
  - Gemeinschaftspraxis am Angerbrunnen, Zwiesel
- Italy (104):
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti
  - P.O. Agrigento Ospedale San Giovanni di Dio, Agrigento
  - IRCCS-INRCA Ancona, Ancona
  - Ospedale di Anzio, Anzio
  - Ospedale dei Castelli, Ariccia
  - Ospedale "C. e G. Mazzoni", Ascoli Piceno
  - A.O. San Giuseppe Moscati, Avellino
  - Ospedale SS Nicola e Filippo, Avezzano
  - Ospedale S. Paolo, Bari
  - A.O.U. Consorziale - Policlinico Bari, Bari
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari - Site 08016, Bari
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari - Site 08017, Bari
  - AUSL Bologna Ospedale di Bentivoglio, Bentivoglio
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna
  - Policlinico Sant'Orsola Bologna-Malpighi, Bologna
  - Ospedale di Bolzano - Site 08070, Bolzano
  - Ospedale di Bolzano - Site 08112, Bolzano
  - Spedali Civili di Brescia, Brescia
  - Ospedale Santo Spirito Casale Monferrato, Casale Monferrato
  - A.O. S. Anna e S. Sebastiano, Caserta
  - ULLS 2 MARCA TREVIGIANA Ospedale di Castelfranco Veneto, Castelfranco Veneto
  - AOU Policlinico Vittorio Emanuele Presidio Ospedaliero Gaspare Rodolico, Catania
  - Azienda Ospedaliera Cannizzaro, Catania
  - L'Azienda Ospedaliero-Universitaria "Renato Dulbecco" di Catanzaro, Catanzaro
  - Ospedale Civile Santa Maria Incoronata dell'Olmo, Cava de' Tirreni
  - Policlinico SS. Annunziata, Chieti
  - ASL TO4 Presidio Riunito di Ciriè-Lanzo, Cirié
  - Azienda Ospedaliero-Universitaria di Ferrara "Arcispedale Sant'Anna", Cona
  - Ospedale San Salvatore, Coppito
  - Ospedale Santa Maria Nuova, Florence
  - AOU Careggi - Site 08067, Florence
  - AOU Careggi - Site 08081, Florence
  - AOU Careggi - Site 08090, Florence
  - Azienda Ospedaliera Universitaria "Ospedali Riuniti" di Foggia, Foggia
  - Ospedale Policlinico San Martino, Genova
  - Presidio Ospedaliero S.O. Padre Antero Micone, Genova
  - Ospedale della Misericordia, Grosseto
  - Ospedale Sant'Andrea, La Spezia
  - ASP Catanzaro Presidio Ospedaliero "Giovanni Paolo II", Lamezia Terme
  - Ospedale Vito Fazzi, Lecce
  - Ospedale Mater Salutis, Legnago
  - Presidio Ospedaliero "Madonna delle Grazie", Matera
  - Presidio ospedaliero San Giovanni di Dio, Melfi
  - A.O.U. Policlinico "G. Martino", Messina
  - ULSS 3 SERENISSIMA Ospedale dell'Angelo, Mestre
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Site 08039, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Site 08097, Milan
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Luca - Gruppo Istituto Auxologico Italiano, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Niguarda, Milan
  - ULSS 3 Serenissima Presidio Ospedaliero di Mirano, Mirano
  - AOU Modena Policlinico Modena, Modena
  - A.O.R.N. Antonio Cardarelli, Napoli
  - A.O.R.N. MONALDI OSPEDALE DEI COLLI Ospedale Monaldi, Napoli
  - A.O.U. Federico Ii, Napoli
  - Azienda Ospedaliera Specialistica dei Colli Ospedale Monaldi, Napoli
  - Policlinico Università Federico II - Napoli, Napoli
  - Ospedale Umberto I, Nocera Inferiore
  - AOU Maggiore della Carità di Novara, Novara
  - Ospedale San Giacomo, Novi Ligure
  - Azienda ospedaliera-Università di Padova, Padua
  - A.O.U. Policlinico "P. Giaccone", Palermo
  - Casa di Cura Triolo Zancla Hospital, Palermo
  - ICS Maugeri, Pavia
  - USL Umbria I, Perugia
  - Azienda Ospedaliera S. Maria della Misericordia di Perugia, Perugia
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Fondazione Monasterio, Pisa
  - P. O. Portogruaro, Portogruaro
  - Azienda Ospedaliera Regionale San Carlo di Potenza, Potenza
  - Nuovo Ospedale Santo Stefano, Prato
  - Azienda Sanitaria Provinciale di Ragusa Ospedale Giovanni Paolo II, Ragusa
  - Ospedale Santa Maria delle Croci, Ravenna
  - ASST Rhodense - Ospedale di Circolo di Rho, Rho
  - Ospedale San Camillo De Lellis, Rieti
  - Ospedale Infermi AUSL Romagna, Rimini
  - Ospedale degli Infermi di Rivoli, Rivoli
  - Policlinico Tor Vergata, Roma
  - Ospedale Sandro Pertini, Roma
  - Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Site 08046, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Site 08121, Roma
  - Policlinico Casilino, Roma
  - AOU S. Andrea, Roma
  - A.O. San Giovanni di Dio e Ruggi D'Aragona, Salerno
  - ASST Valle Olona P.O. Saronno, Saronno
  - Ospedale S. Bartolomeo, Sarzana
  - AOU Sassari Ospedale SS. Annunziata, Sassari
  - IRCCS Multimedica, Sesto San Giovanni
  - A.O.U. Senese Ospedale Santa Maria alle Scotte, Siena
  - AOU Senese- Policlinico Le Scotte, Siena
  - Casa di cura Villa Verde, Taranto
  - Azienda Ospedaliera Santa Maria, Terni
  - Ospedale Mauriziano Presidio Umberto I, Torino
  - AOU Ospedali Riuniti di Ancona, Torrette
  - Ospedale Santa Chiara, Trento
  - ULLS 2 MARCA TREVIGIANA Ospedale Ca' Foncello, Treviso
  - Ospedale di Cattinara, Trieste
  - Ospedale Santa Maria della Misericordia, Udine
  - Ospedale Santa Maria della Misericordia, Urbino
  - ASST Settelaghi Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Castelli Verbania, Verbania
- Netherlands (21):
  - ZGT, Almelo
  - Meander Mc, Amersfoort
  - AUMC, Amsterdam
  - Mc Leeuwarden, Amsterdam
  - Rijnstate, Arnhem
  - AMPHIA, Breda
  - Albert Schweitzer, Dordrecht
  - ZGV, Ede
  - Maxima Medisch Centrum, Eindhoven
  - GHZ, Gouda
  - Spaarne Gasthuis, Haarlem
  - Saxenburgh Medisch Centrum, Hardenberg
  - Tergooi Mc, Hilversum
  - Treant Bethesda Hoogeveen, Hoogeveen
  - Dijklander, Hoorn
  - ALRIJNE, Leiderdorp
  - MUMC+, Maastricht
  - Erasmus Mc, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - MAASSTAD, Rotterdam
  - Isala Zwolle, Zwolle
- Spain (68):
  - Hospital General de Albacete, Albacete
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Hospital Virgen de los Lirios, Alcoy
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Universitario Central de Asturias, Asturias
  - Clínica Mapfre Salud Gijón, Asturias
  - Hospital Universitario San Agustin, Asturias
  - Hospital Vital Álvarez-Buylla, Asturias
  - Hospital Universitario Nuestra Señora del Perpetuo Socorro, Badajoz
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital de Bellvitge, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario de Castellón, Castellon
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital del Henares, Coslada, Madrid
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital de Denia, Denia
  - Hospital UNiversitario de Donostia, Donostia / San Sebastian
  - Hospital de Fuenlabrada, Fuenlabrada Madrid
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Médico-Quirúrgico de Jaén, Jaén
  - Hospital Jerez de la Frontera, Jerez de La Frontera, Cádiz
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Complejo Hospitalario Universitario Insular Materno-Infantil de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital San Pedro, Logroño
  - Hospital Universitario la Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital HM Montepríncipe, Madrid
  - Hospital Universitario de Torrejón, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majdahonda Madrid
  - Hospital Costa del Sol, Marbella Málaga
  - Consulta de Cardiología Dr. Javier Mora Robles, Málaga
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital de Mendaro, Mendaro
  - Hospital General Universitario Reina Sofía, Murcia
  - Hospital Clínico Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Son LLatzer, Palma de Mallorca
  - Hospital Universitario de Navarra, Pamplona
  - Hospital de Sagunto, Port de Sagunt
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital de Valme, Seville
  - Hospital Universitario Vírgen del Rocío, Seville
  - Hospital General Universitario de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Vithas Valencia 9 de Octubre, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital de La Plana, Villarreal, Castellón
  - Hospital Clinico Universitaro Lozano Blesa, Zaragoza
- Switzerland (17):
  - Diabetologie & Endokrinologie Baden, Baden
  - University Hospital Basel, Basel
  - Inselspital, Universitätsspital Bern, Bern
  - Praxis Dr. med Urs Beat Gröflin, Binningen
  - Hochgebirgsklinik Davos, Davos
  - Spital Lachen AG, Lachen
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - University of Lausanne, Lausanne
  - Kantonsspital Baselland, Liestal
  - EOC Ente Ospedaliero Cantonale, Lugano
  - MIP Associazione Medico in Pratica c/o Studio Medico Cardiologico Acquistapace, Lugano
  - Praxis Prof. Dr. med. Gottfried Rudofsky, Olten
  - HÔPITAL RIVIERA-CHABLAIS, VAUD-VALAIS, Centre hospitalier de Rennaz, Rennaz
  - Kantonsspital St.Gallen, Sankt Gallen
  - Spital Thun, Thun
  - Prof. Dr. med. Stephane Bosquet, Yverdon-les-Bains
  - Universitätsspital Zürich, Zurich
- United Kingdom (31):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - South Eastern Ulster Hospital, Belfast
  - University Hospital of Wales, Cardiff
  - Rowden Surgery, Chippenham
  - Craigavon Area Hospital, Craigavon
  - Darlington Memorial Hospital, Darlington
  - University Hospital North Durham, Durham
  - Oaks Healthcare, Hampshire
  - West Morland General Hospital, Kendal
  - North Blaby PCN, Leicester
  - Barts Health NHS Trust/ QMUL, London
  - Freuchen Medical Centre, London
  - Royal Free Hospital Lipid Clinic, London
  - Hammersmith Hospital, London
  - Imperial College London, London
  - Manchester Royal Infirmary, Manchester
  - Manchester University NHS Foundation Trust, Manchester
  - Wythenshawe Hospital, Manchester
  - STRIVE, The James Cook University Hospital, Middlesbrough
  - North Tees Hospital, Northumbria
  - City Hospital, Nottingham
  - Queen Alexandra Hospital, Portsmouth
  - Whiston Hospital, Prescot
  - North Manchester General Hospital, Salford
  - Queen's Hospital Lipid Clinic, Staffordshire
  - Princess Royal Hospital, Telford
  - Torbay and South Devon NHS Foundation Trust, Torquay
  - Trowbridge Health Centre, Trowbridge
  - North Wales Cardiac Centre, Wales
  - Wansford and Kings Cliffe Practice, Wansford
  - Bridgewater Surgeries, Watford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/